CLINICAL TRIAL: NCT00536731
Title: A 6-week, Phase III, Double-blind, Randomized, Multi-centre, Parallel-group Study Evaluating the Efficacy and Safety of 2 Actuations Symbicort®pMDI® 40/2.25 μg Twice Daily Compared With 1 Inhalation Symbicort Turbuhaler® 80/4.5 μg Twice Daily and 1 Inhalation Pulmicort®Turbuhaler® 100 μg Twice Daily
Brief Title: Symbicort Rapihaler Therapeutic Equivalence Study
Acronym: ESTHER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5897C00003
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Results first posted 2012-08-15 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Bronchial Asthma
Keywords: Asthma; Symbicort
MeSH Terms: conditions — Asthma | interventions — Budesonide, Formoterol Fumarate Drug Combination; Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Symbicort pMDI (Active Comparator): Symbicort®pMDI® 40/2.25 μg 2 Actuations Twice Daily
  Interventions: Drug: Symbicort pMDI
- Symbicort Turbuhaler (Active Comparator): Symbicort Turbuhaler® 80/4.5 μg 1 Inhalation Twice Daily
  Interventions: Drug: Symbicort Turbuhaler
- Pulmicort Turbuhaler (Active Comparator): Pulmicort®Turbuhaler® 100 μg 1 Inhalation Twice Daily
  Interventions: Drug: Pulmicort Turbuhaler

INTERVENTIONS:
Drug: Symbicort Turbuhaler — Symbicort Turbuhaler® 80/4.5 μg 1 Inhalation Twice Daily
  Arms: Symbicort Turbuhaler
Drug: Symbicort pMDI — Symbicort®pMDI® 40/2.25 μg 2 Actuations Twice Daily
  Arms: Symbicort pMDI
Drug: Pulmicort Turbuhaler — Pulmicort®Turbuhaler® 100 μg 1 Inhalation Twice Daily
  Arms: Pulmicort Turbuhaler

SUMMARY:
The purpose of the this study is to evaluate the efficacy and safety of 2 actuations Symbicort®pMDI® 40/2.25 μg twice daily compared with1 inhalation Symbicort Turbuhaler® 80/4.5 μg twice daily and 1 inhalation Pulmicort®Turbuhaler® 100 μg twice daily for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Asthma clinically diagnosed since at least 6 months.
* Lung function values measured ≥ 50% and ≤ 90% of predicted normal.
* Patients with reversible airway obstruction Daily use of inhaled steroids (any brand) for >3 months.

Exclusion Criteria:

* Use of oral, rectal or parenteral steroids within 30 days prior to start of study.
* Respiratory infection affecting the asthma, as judged by the investigator, within 30 days prior to start of randomised treatment.
* Any significant disease or disorder which, in the opinion of the investigator, may either put the patient at risk because of participation in the study, or may influence the results of the study or the patient's ability to participate in the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 742 (Actual)
Dates: Start 2007-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Andersson, Study Director — AstraZeneca; Akos Somoskovi, Principal Investigator — AstraZeneca
Locations (48):
- Bulgaria (5):
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Varna
- Czechia (12):
  - Research Site, Benesov U Prahy
  - Research Site, Hradec Králové
  - Research Site, Jihlava
  - Research Site, Kladno
  - Research Site, Kolín
  - Research Site, Kutná Hora
  - Research Site, Litoměřice
  - Research Site, Neratovice
  - Research Site, Pardubice
  - Research Site, Prague
  - Research Site, Rokycany
  - Research Site, Strakonice
- Hungary (13):
  - Research Site, Balassagyarmat
  - Research Site, Budapest
  - Research Site, Cegléd
  - Research Site, Debrecen
  - Research Site, Deszk
  - Research Site, Győr
  - Research Site, Gyula
  - Research Site, Kaposvár
  - Research Site, Nyíregyháza
  - Research Site, Szarvas
  - Research Site, Százhalombatta
  - Research Site, Szeged
  - Research Site, Törökbálint
- Poland (18):
  - Research Site, Bialystok
  - Research Site, Bielsko-Biala
  - Research Site, Bydgoszcz
  - Research Site, Chodzież
  - Research Site, Chrzanów
  - Research Site, Karpacz
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Ostrów Wielkopolski
  - Research Site, Poznan
  - Research Site, Skierniewice
  - Research Site, Szczecin
  - Research Site, Tarnów
  - Research Site, Turek
  - Research Site, Wodzisław Śląski
  - Research Site, Wroclaw
  - Research Site, Łomża

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 898 subjects enrolled; 156 not randomised: 94 incorrect enrolment, 9 adverse events, 18 voluntary discontinuations, 1 lost to follow-up, 1use of not allowed medication, 1 non-compliant
Period: Overall Study
Arm/Group | Symbicort pMDI | Symbicort Turbuhaler | Pulmicort Turbuhaler
Started | 253 | 246 | 243
Completed | 249 | 241 | 238
Not Completed | 4 | 5 | 5
Not completed — Adverse Event | 3 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — Intake of prohibited conc. medication | 0 | 0 | 1
Not completed — Safety reasons | 0 | 0 | 1
Not completed — Other | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Symbicort pMDI | Symbicort Turbuhaler | Pulmicort Turbuhaler | Total
Number analyzed (Participants) | 253 | 246 | 243 | 742
Age Continuous [Mean (Full Range); unit: years] | 41 [12 to 75] | 42 [12 to 76] | 39 [12 to 78] | 41 [12 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 142 | 131 | 425
  Male | 101 | 104 | 112 | 317

OUTCOME MEASURES:

1. Primary Outcome: Morning Peak Expiratory Flow (PEF)
Description: Change in the Morning PEF from baseline (calculated as a mean using all available data for the 10 last days of run-in period) to week 6 (calculated as a mean using all available data after randomisation). No imputation of missing data was performed
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: Liters/min
Arm/Group | Symbicort pMDI | Symbicort Turbuhaler | Pulmicort Turbuhaler
Number analyzed (Participants) | 253 | 245 | 243
Liters/min | 12.88 (24.6) | 13.78 (29.7) | 4.59 (27.9)

2. Secondary Outcome: Evening Peak Expiratory Flow (PEF)
Description: Change in the Evening PEF from baseline (calculated as a mean using all available data for the 10 last days of run-in period) to week 6 (calculated as a mean using all available data after randomisation). No imputation of missing data was performed
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: Liters/min
Arm/Group | Symbicort pMDI | Symbicort Turbuhaler | Pulmicort Turbuhaler
Number analyzed (Participants) | 253 | 245 | 243
Liters/min | 12.34 (24.3) | 10.80 (29.1) | 1.43 (25.7)

3. Secondary Outcome: Asthma Symptom Score, Night
Description: Change in the Asthma Symptom Score (Night) from baseline (calculated as a mean using all available data for the 10 last days of run-in period) to week 6 (calculated as a mean using all available data after randomization, with run-in values as covariate). No imputation of missing data was performed. Daily scale:0 = No symptoms; 1 = Mild symptoms; 2 = Moderate symptoms; 3 = Severe symptoms.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Symbicort pMDI | Symbicort Turbuhaler | Pulmicort Turbuhaler
Number analyzed (Participants) | 253 | 245 | 243
Units on a scale | -0.24 (0.41) | -0.27 (0.41) | -0.15 (0.39)

4. Secondary Outcome: Asthma Symptom Score, Day
Description: Change in the Asthma Symptom Score (Day) from baseline (calculated as a mean using all available data for the 10 last days of run-in period) to week 6 (calculated as a mean using all available data after randomization, with run-in values as covariate). No imputation of missing data was performed. Daily scale:0 = No symptoms; 1 = Mild symptoms; 2 = Moderate symptoms; 3 = Severe symptoms.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Symbicort pMDI | Symbicort Turbuhaler | Pulmicort Turbuhaler
Number analyzed (Participants) | 253 | 245 | 243
Units on a scale | -0.21 (0.38) | -0.24 (0.40) | -0.15 (0.40)

5. Secondary Outcome: Asthma Symptom Score, Total
Description: Change in the Asthma Symptom Score (Total) from baseline (calculated as a mean using all available data for the 10 last days of run-in period) to week 6 (calculated as a mean using all available data after randomization, with run-in values as covariate). No imputation of missing data was performed. Daily scale:0 = No symptoms; 1 = Mild symptoms; 2 = Moderate symptoms; 3 = Severe symptoms.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Symbicort pMDI | Symbicort Turbuhaler | Pulmicort Turbuhaler
Number analyzed (Participants) | 253 | 245 | 243
Units on a scale | -0.45 (0.73) | -0.51 (0.75) | -0.30 (0.73)

6. Secondary Outcome: Percentage of Nights With Awakenings Due to Asthma
Description: Change in the Percentage of Nights With Awakenings Due to Asthma from baseline (calculated as a mean using all available data for the 10 last days of run-in period) to week 6 (calculated as a mean using all available data after randomization, with run-in values as covariate). No imputation of missing data was performed. The participants answered "Yes" or "No" whether she/he woke up during the night due to asthma.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: Percentage of night
Arm/Group | Symbicort pMDI | Symbicort Turbuhaler | Pulmicort Turbuhaler
Number analyzed (Participants) | 253 | 245 | 243
Percentage of night | -14.0 (24.1) | -14.0 (26.4) | -8.3 (25.5)

7. Secondary Outcome: Use of Rescue Medication, Night
Description: Change in the Use of Rescue Medication (Night) from baseline (calculated as a mean using all available data for the 10 last days of run-in period) to week 6 (calculated as a mean using all available data after randomization, with run-in values as covariate). No imputation of missing data was performed
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: Inhalations
Arm/Group | Symbicort pMDI | Symbicort Turbuhaler | Pulmicort Turbuhaler
Number analyzed (Participants) | 253 | 245 | 243
Inhalations | -0.41 (0.64) | -0.39 (0.76) | -0.19 (0.67)

8. Secondary Outcome: Use of Rescue Medication, Day
Description: Change in the Use of Rescue Medication (Day) from baseline (calculated as a mean using all available data for the 10 last days of run-in period) to week 6 (calculated as a mean using all available data after randomization, with run-in values as covariate). No imputation of missing data was performed
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: Inhalations
Arm/Group | Symbicort pMDI | Symbicort Turbuhaler | Pulmicort Turbuhaler
Number analyzed (Participants) | 253 | 245 | 243
Inhalations | -0.21 (0.39) | -0.20 (0.47) | -0.13 (0.56)

9. Secondary Outcome: Use of Rescue Medication, Total
Description: Change in the Use of Rescue Medication (Total) from baseline (calculated as a mean using all available data for the 10 last days of run-in period) to week 6 (calculated as a mean using all available data after randomization, with run-in values as covariate). No imputation of missing data was performed
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: Inhalations
Arm/Group | Symbicort pMDI | Symbicort Turbuhaler | Pulmicort Turbuhaler
Number analyzed (Participants) | 253 | 245 | 243
Inhalations | -0.62 (0.89) | -0.58 (1.09) | -0.32 (1.12)

10. Secondary Outcome: Percentage of Symptom-free Days
Description: Change in the Percentage of Symptom-free Days from baseline (calculated as a mean using all available data for the 10 last days of run-in period) to week 6 (calculated as a mean using all available data after randomization, with run-in values as covariate). No imputation of missing data was performed. Symptom-free Day: no symptoms (asthma symptom score=0) night and day, and no awakenings due to asthma.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Symbicort pMDI | Symbicort Turbuhaler | Pulmicort Turbuhaler
Number analyzed (Participants) | 253 | 245 | 243
Percentage of days | 12.5 (23.7) | 15.3 (24.5) | 9.1 (21.2)

11. Secondary Outcome: Percentage of Asthma Control Days
Description: Change in the Percentage of Symptom Control Days from baseline (calculated as a mean using all available data for the 10 last days of run-in period) to week 6 (calculated as a mean using all available data after randomization, with run-in values as covariate). No imputation of missing data was performed. Asthma Control Day: no symptoms (asthma symptom score=0) night and day, no awakenings due to asthma, no rescue medication.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Symbicort pMDI | Symbicort Turbuhaler | Pulmicort Turbuhaler
Number analyzed (Participants) | 253 | 245 | 243
Percentage of days | 12.7 (23.6) | 15.1 (24.4) | 9.1 (21.2)

12. Secondary Outcome: Percentage of Rescue Free Days
Description: Change in the Percentage of Rescue Free Days from baseline (calculated as a mean using all available data for the 10 last days of run-in period) to week 6 (calculated as a mean using all available data after randomization, with run-in values as covariate). No imputation of missing data was performed. Rescue-free Day defined as day and night with no use of rescue medication.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Symbicort pMDI | Symbicort Turbuhaler | Pulmicort Turbuhaler
Number analyzed (Participants) | 253 | 245 | 243
Percentage of days | 24.0 (30.9) | 26.2 (30.7) | 17.2 (28.4)

13. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1)
Description: Change in the FEV1from baseline to week 6 (calculated as a mean using all available data after randomization)
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort pMDI | Symbicort Turbuhaler | Pulmicort Turbuhaler
Number analyzed (Participants) | 253 | 243 | 242
Liters | 0.095 (0.328) | 0.147 (0.364) | 0.112 (0.326)

ADVERSE EVENTS:
Groups:
- Symbicort pMDI: Symbicort pMDI
- Symbicort Turbuhaler: Symbicort Turbuhaler
- Pulmicort Turbuhaler: Pulmicort Turbuhaler
Arm/Group | Symbicort pMDI | Symbicort Turbuhaler | Pulmicort Turbuhaler
Serious Adverse Events (participants affected / at risk) | 0/253 | 1/246 | 1/243
Other Adverse Events (participants affected / at risk) | 0/253 | 0/246 | 0/243
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Symbicort pMDI (N=253) | Symbicort Turbuhaler (N=246) | Pulmicort Turbuhaler (N=243)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No